CLINICAL TRIAL: NCT05892484
Title: High Resolution Infrared Thermography as a Diagnostic Aid in Paediatric Wrist Injuries Version 2
Brief Title: HiRes Infrared Imaging for Wrist Injuries in Children v2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SCH-2323
Record Dates: First submitted 2021-06-04; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone | interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: Comparison between thermal imaging and x-ray.
Who Masked: Care Provider
Masking Description: If the thermal imaging is done first, the radiographer taking the x-ray won't be informed of the outcome of the imaging assessment, so two independent assessments can be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thermal Imaging (Experimental): Participants will receive thermal imaging in addition to their routine x-ray for comparison.
  Interventions: Device: Thermal Imaging
- X-ray (Other): Routine x-ray is what the active comparator is being evaluated against.
  Interventions: Diagnostic Test: X-RAY

INTERVENTIONS:
Device: Thermal Imaging — Thermal Imaging device used to evaluate fracture in those presenting with proposed wrist fracture in the emergency department.
  Arms: Thermal Imaging
Diagnostic Test: X-RAY — Routine X-RAY
  Arms: X-ray

SUMMARY:
When assessing an injured child, doctors must decide whether or not there is an underlying bony fracture. The current way of doing this is by x-ray. In 2011, 46,000 children attended Sheffield Children's Hospital Emergency Department and 10,400 x-rays were taken - predominately for diagnosis of fractures. For foot and wrist, 2,215 x-rays were 'normal' with no fracture, at a cost of £119,610 (at a tariff of £54 per x-ray). Considering the cost and undesired effect of radiation exposure, a better way to discriminate those patients with fracture is needed. The non-invasive technique of thermal imaging holds promise as a putative technique.

The investigators have earlier demonstrated the potential of thermal imaging for vertebral fractures, diagnosing limp and measuring respiration rate. This study investigates thermal imaging to screen for wrist fractures. The objectives are: (i) accurately identify fracture location, (ii) exclude cases that are sprain and thus reduce the need for their x-ray. The confirmation of a fracture would still require a x-ray. As the study is in collaboration with Sheffield Children's Hospital, only children will be included, however the findings will also be applicable to adults. Thermal imaging is a completely safe and harmless operation, as the camera is non-contact and emits no radiation.

Any trauma, such as a wrist fracture, results in changes in blood flow that in turn affects the skin surface temperature of the skin overlying the injury. These changes affect the amount of emitted infrared radiation and will be recorded and explored to find a marker to differentiate fractures and sprains.

DETAILED DESCRIPTION:
Thermal (IR) imaging is based on recording and processing of a part of electromagnetic spectrum below visible light, i.e. infrared band. Objects with a temperature above -273°C (- 459.67°F) emit thermal radiation. In thermography a camera that is sensitive to the mid (3-5 μm) and long (7-14 μm) infrared bands of the electromagnetic spectrum is used. The detection of an injury using thermal imaging relies on underlying physiology of temperature differentials.

Dermal temperature differentials usually do not exceed 0.25°C, while differentials in excess of 0.65°C are consistently related to pathology. Therefore observation of a significant temperature differential is an indication of injury. The use of Infrared for musculoskeletal medical diagnosis and monitoring has been reported in many studies in children and adults.

* Vertebral fractures were detected using thermal imaging • Thermal imaging assisted in diagnosis of the causes of limp including bone fracture.

Thermography has detected a direct correlation between an increase in skin temperature and the existence of anterior) knee pain after implantation of artificial knee joints. It is suggested that thermal imaging is potentially valuable for a rapid, inexpensive and non-invasive diagnosis of pain and inflammation. Infrared spectroscopic analysis has been reported to be is a powerful tool for establishing the material properties that contribute to bone strength and so it thus has been helpful in improving the understanding of the changes in fragile bone.

• The temperature of the bone during drilling could increase above 47oC. This can cause irreversible osteonecrosis. A study used infrared thermal imaging to determine spatial distribution of increase in bone temperature during drilling.

Blood convection warms the skin by transfer of heat from the core and this process plays the major role in determining skin temperature. Skin's has a thermoregulation role, i.e. it generates, absorbs, conducts and radiates heat. Changes in the skin surface temperature are valuable in detecting physiological and pathological state such as inflammation.

With recent developments in thermal imaging devices, the use of infrared imaging for injury examination is gaining a growing interest, with more evidence supporting its use. However, the data in children is limited, with the investigators' research group undertaking the majority of work in this field currently.

In this study the infrared emission (characterised by heat radiation) from skin at the site of injury is imaged and analysed to differentiate between wrist fracture and sprain. The hypothesis is that the inflammation and blood perfusion in sprain and bone fracture at the site of injury are different leading to distinct temperature gradients at the site.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-16 years who are admitted to the Emergency Department of Sheffield Children's Hospital for a wrist injury, and who are x-rayed as part of their standard clinical management. Inclusion is subject to both the patient and carer having read (or being read to in very young children) the information sheets and both the patient and carer consenting to participate.

Exclusion Criteria:

* Children who have multiple injuries (e.g. those involved in serious car accident accidents).
* Children who are too distressed (by pain or otherwise).
* Parents/carers who have difficulty understanding the nature of the study (e.g. non-native English speakers, those with disabilities impairing their understanding of the study etc.) will be excluded.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
The Accuracy of Thermal Imaging to Detect Fractures | 12 months
  Percentage of fractures correctly identified by Thermal Imaging.
Diagnostic accuracy of Thermal Imaging | 12 months
  Sensitivity and Specificity of thermal imaging in identifying or excluding fractures

CONTACTS AND LOCATIONS:
Overall Officials: Shammi Ramlakhan, Principal Investigator — Sheffield Children's NHS Trust
Locations (1):
- Clinical Research Facility, Sheffield Children's Hospital, Sheffield, United Kingdom